CLINICAL TRIAL: NCT04896021
Title: Improved Cardiovascular Disease hEALth Service Delivery in Australia: Cluster Randomised Controlled Trial (IDEAL Study)
Acronym: IDEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menzies Institute for Medical Research (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Diagnostic Services Pty Ltd (Unknown); Department of Health, Tasmania (Other Government); Primary Health Tasmania (Unknown); National Heart Foundation, Australia (Other); Healthcare Software Pty Ltd (Unknown); Uscom Limited (Unknown)
Responsible Party: Principal Investigator, james E sharman, Professor, Menzies Institute for Medical Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HREC23015; GNT1170815 (Other Grant/Funding Number: NHMRC)
Record Dates: First submitted 2021-05-11; First posted 2021-05-21 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular disease risk management
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Participants attending pathology services for blood cholesterol assessment will be randomized to intervention or control arms. Randomization is clustered at the level of general practice clinics (n=60 target) referring patients to pathology services for blood cholesterol assessment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Allocation is concealed from all people involved in eligibility screening and recruitment.
  Pathology services reception and blood collection staff members may be employed across different collection centers that could include both intervention and control sites. Thus, concealment at the cluster level (as per this study design) is critical and all procedures undertaken by staff members interacting with participants (reception and blood collection staff) will be identical. At the participant level, there will be no indication provided regarding allocation (all participants will have the same information and undergo the same protocol at baseline assessment). Investigators will be blinded to participant allocation. Outcomes assessment is via linkage to health outcomes data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): On referral to Tasmanian pathology services for blood cholesterol, intervention participants will have their blood pressure measured and collated with other cardiovascular disease risk factors. An absolute cardiovascular disease risk score is calculated, interpreted according to guideline recommendations and reported to referring doctors via the established pathology system. High risk is highlighted in red as per usual practice for pathology tests outside of normal range, and advice provided regarding appropriate action according to National Vascular Disease Prevention Alliance guidelines.
  Interventions: Diagnostic Test: Cardiovascular disease risk assessment
- Control (Active Comparator): On referral to Tasmanian pathology services for blood cholesterol, control participants will have their blood pressure measured and collated with other cardiovascular disease risk factors as per the intervention arm. However, only the results relating to blood cholesterol are reported to the referring doctor, as per usual practice.
  Interventions: Diagnostic Test: Usual care assessment

INTERVENTIONS:
Diagnostic Test: Cardiovascular disease risk assessment — Intervention in which the addition of guideline-recommended absolute cardiovascular disease risk assessment is embedded into point-of-care blood collection services for cholesterol measurement and results (including risk score) are reported to referring doctors.
  Arms: Intervention
Diagnostic Test: Usual care assessment — Usual care in which blood cholesterol results are reported to referring doctors
  Arms: Control

SUMMARY:
The IDEAL study is a randomized controlled trial among people referred to pathology services to have blood cholesterol measured. Study participants will have cardiovascular risk factors (e.g. age, sex, blood pressure, diabetes, smoking status) measured within an assessment station at pathology services. A report on cardiovascular risk, in addition to blood cholesterol results, will be sent to the referring doctor along with recommended treatment strategies among those participants randomized to intervention. For control participants, the usual care process will be provided in which only blood cholesterol results will be sent to the referring doctor. The new intervention is expected to lead to better identification and treatment of people at high risk for cardiovascular disease events.

DETAILED DESCRIPTION:
The IDEAL study aims to improve the way doctors identify and manage patients at risk of cardiovascular disease, including conditions such as heart attack or stroke. This research focuses on an improved service to work out a patient's risk of heart attack or stroke and deliver this information to doctors to help them make well-informed treatment decisions to prevent cardiovascular disease and improve outcomes for their patients.

This IDEAL study is a randomized clinical trial of the IDEAL service to be conducted among 9,714 participants attending pathology services in Tasmania, Australia.

Patients attending pathology service clinics around Tasmania for a cholesterol test may be invited to participate. Participants will have their risk of cardiovascular disease assessed in a purpose-built assessment station where information about their cardiovascular disease risk factors, such as smoking, will be collected and blood pressure measured. An estimate of the chances of that patient having a heart attack or stroke in the next 5 years will be calculated and sent to their referring doctor along with their pathology results on the requested blood test report.

Based on the patient's risk of cardiovascular disease, appropriate advice according to recommended treatment guidelines will be provided on the pathology report as an aid for doctors to make better-informed decisions to manage patients at risk of cardiovascular disease.

Participants will also be asked to complete a questionnaire to explore issues of cardiovascular disease risk in more depth, with follow-up questionnaires at 6 and 12 months. After 12 months researchers will examine if there is an improvement in cardiovascular disease risk management and health outcomes for participants whose doctors received the cardiovascular disease risk information on the pathology report. This will be done through data linkage with national and state level data, as well as through asking participants to re-complete the questionnaire.

In addition, a qualitative research program will be conducted to understand the barriers and enablers to uptake of the IDEAL service from the perspective of pathology staff, doctors and patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to pathology services for blood cholesterol (lipids; total cholesterol and HDL cholesterol) who are eligible for absolute CVD risk assessment according to the National Vascular Disease Prevention Alliance guidelines (this includes all adults aged 45 years and over without a known history of CVD, or Aboriginal and Torres Strait Islander people aged 35 years or over) and willing to provide permission to access to PBS-linked data on medications prescribed and dispensed.
* Adults already deemed to be at increased risk that do not require absolute CVD risk assessment according to guidelines will also be included because there is evidence that these people are undertreated (Heeley EL, et al Med J Aust 2010;192:254-9; Peiris DP, et al Med J Aust 2009;191:304-9) and therefore may benefit from improved assessment. This includes adults with any of the following: Diabetes and age >60 years; Diabetes with microalbuminuria (>20 mcg/min or urinary albumin:creatinine ratio >2.5 mg/mmol for males, >3.5 mg/mmol for females); Moderate or severe CKD (persistent proteinuria or estimated glomerular filtration rate (eGFR) <45 mL/min/1.73 m2); A previous diagnosis of familial hypercholesterolaemia; Serum total cholesterol >7.5 mmol/L; Aboriginal and Torres Strait Islander adults aged over 74

Exclusion Criteria:

* Adults already taking antihypertensive or lipid lowering medications (determined by self-report at baseline)
* if the referring doctor is not from a general practice included in the study cluster list,
* if participants cannot provide an email address to be used to provide a copy of their signed consent form.
* If at least one measurement of blood pressure is unable to be obtained at baseline assessment.
* For safety reasons, people will be excluded if they are found at the time of assessment at the pathology services with an average systolic blood pressure =180 mmHg or diastolic blood pressure =110 mmHg.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2761 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Antihypertensive and/or statin medications dispensed | 1 year after randomization
  Antihypertensive and/or statin medications dispensed, confirmed by data linkage to Pharmaceutical Benefits Scheme

SECONDARY OUTCOMES:
Cost effectiveness | 1 year after randomization
  Cost effectiveness of intervention compared with usual care
Barriers and enablers | 1 year after randomization
  Barriers and enablers to implementation and uptake of intervention as ascertained from pathology services staff, referring doctors and patients

OTHER OUTCOMES:
Cardiovascular outcomes | This tertiary-level exploratory analysis will be conducted to determine power for future trials. Analysis will be performed after accrual of events that are anticipated to occur after at least 2 years follow-up
  Cardiovascular-related hospitalizations, procedures and events, including mortality, ascertained via data linkage

CONTACTS AND LOCATIONS:
Overall Officials: James E Sharman, PhD, Principal Investigator — Menzies Institute for Medical Research
Locations (1):
- Menzies Institute for Medical Research, Hobart, Tasmania, Australia

IPD SHARING:
Plan to Share IPD: Yes
The deidentified study data, including data dictionaries, will be made publicly available on reasonable request via the University of Tasmania's Research Data Portal (consistent with the Australian Code for the Responsible Conduct of Research).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after publication of the principal findings
Access Criteria: Access subject to approvals by the Principal Investigator consistent with the Australian Code for the Responsible Conduct of Research.

REFERENCES:
- [Derived] Pagano L, Sharman JE, Nash R, Sutton L, Donovan S, Owens D, Murfett L, Heathcote S, Wells G, Zurynski Y, Sarkies M, Chapman N. Implementing absolute cardiovascular disease risk assessment into pathology collection services. J Eval Clin Pract. 2024 Oct;30(7):1239-1250. doi: 10.1111/jep.14034. Epub 2024 Jun 3. PMID 38828679